CLINICAL TRIAL: NCT00004180
Title: Phase II Clinical Trial of Rosiglitazone, a Full-Agonist Ligand for the Peroxisome Proliferator-Activated Receptor Gamma (PPAR), as Differentiation Therapy for Patients With Liposarcoma
Brief Title: Rosiglitazone in Treating Patients With Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, George Demetri, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067406; P30CA006516 (NIH); DFCI-99083 (Other: Dana-Farber Cancer Institute); NCI-G99-1629
Record Dates: First submitted 2000-01-21; First posted 2003-05-09 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Sarcoma
Keywords: adult liposarcoma; recurrent adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Liposarcoma | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Well-differentiated liposarcoma (Experimental): Participants in this arm receive 4 mg of study drug (rosiglitazone maleate) twice daily by mouth.
  Interventions: Drug: rosiglitazone maleate
- De-differentiated liposarcoma (Experimental): Participants in this arm receive 4 mg of study drug (rosiglitazone maleate) twice daily by mouth.
  Interventions: Drug: rosiglitazone maleate
- Myxoid/ round-cell liposarcoma (Experimental): Participants in this arm receive 4 mg of study drug (rosiglitazone maleate) twice daily by mouth.
  Interventions: Drug: rosiglitazone maleate
- Pleomorphic liposarcoma (Experimental): Participants in this arm receive 4 mg of study drug (rosiglitazone maleate) twice daily by mouth.
  Interventions: Drug: rosiglitazone maleate

INTERVENTIONS:
Drug: rosiglitazone maleate
  Other Names: Rosiglitazone

SUMMARY:
RATIONALE: Rosiglitazone may help liposarcoma cells develop into normal fat cells.

PURPOSE: Phase II trial to study the effectiveness of rosiglitazone in treating patients who have liposarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical activity of rosiglitazone in patients with liposarcoma.
* Assess the impact of this regimen on markers of tumor proliferation and differentiation status in these patients using biologic and biochemical testing and correlative imaging.
* Determine the tolerance and safety of this regimen in these patients.

OUTLINE: Patients are stratified by histologic subtype (well differentiated vs dedifferentiated vs myxoid/round cell vs pleomorphic).

Patients receive oral rosiglitazone twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1-3 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 56-120 patients (14-30 per stratum) will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven liposarcoma that is incurable with standard multimodality approaches (e.g., surgery and/or radiotherapy and/or chemotherapy)

  * Well differentiated OR
  * Dedifferentiated OR
  * Myxoid/round cell OR
  * Pleomorphic
* Measurable disease
* No clinically unstable brain metastases
* No progression on prior troglitazone therapy for liposarcoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 90,000/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT less than 5 times upper limit of normal

Renal:

* Creatinine no greater than 2.4 mg/dL

Cardiovascular:

* No poorly controlled atrial arrhythmias, symptomatic angina pectoris, or myocardial infarction within the past 4 months
* No symptomatic congestive heart failure, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

  * Oral contraceptives are not considered effective contraception
* No active retroviral disease
* No condition that would preclude informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior chemotherapy allowed and recovered
* No concurrent cytotoxic therapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed and recovered
* At least 6 months since prior radiotherapy to the sole site of measurable disease
* Concurrent localized radiotherapy to a single site of disease allowed if there are other sites of measurable disease

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1999-10; Primary Completion 2006-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evidence of biological response
  Evidence of biological response can be measured or defined by intracytoplasmic microvesicular lipid accumulation, consistent with adipocytic differentiation in liposarcoma cells. Biological response can also be measured by clinically stable disease for x>3 months, as well as standard clinical trial criteria for "objective clinical response." Complete response is defined by total resolution of all detectable disease lasting for at least four weeks. Partial remission is a decrease of over 50% in the sum of the products of the largest perpendicular diameters of all measurable lesions, persisting for at least four weeks, without progression of any non-measurable sites, and without appearance of any new sites of disease.

CONTACTS AND LOCATIONS:
Overall Officials: George D. Demetri, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No